CLINICAL TRIAL: NCT02869685
Title: Consistency Analysis of PD-L1s in Non-small Cell Lung Cancer Patients' Cancer Tissues and in Plasma Exosomes Before and After Radiotherapy:A Clinical Trial
Brief Title: Consistency Analysis of PD-L1s in Advanced NSCLC Tissues and in Plasma Exosomes Before and After Radiotherapy
Acronym: RadImm02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy Director, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-003
Record Dates: First submitted 2016-08-02; First posted 2016-08-17 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: NSCLC
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a prospective, open,phase I clinical study (Other): The investigators have designed five kinds of radiation-division with bioequivalent doses, and detected the expression levels of PD-L1 in pExo after 24h, 48h of each stage of radiotherapy.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy

SUMMARY:
The detection of tissue PD-L1 immunohistochemistry in NSCLC has an important role in guiding for the treatment of immune detection point.Radiation therapy can enhance the effect of immunotherapy,but radiation dose and timing are waiting to be solved. At the same time,tissue detection is time-consuming and laborious, liquid biopsy can reflect the information of tumor tissue,PD-L1 mRNA in plasma exosomes (pExo) is expected to be simple, rapid, non-invasive means of detection. The project is planned to explore the consistency analysis of PD-L1 expression level detected in advanced non-small cell cancer patients' cancer tissues and pExo before and after radiotherapy.The investigators have designed five kinds of radiation-division with bioequivalent doses, and detected the expression levels of PD-L1 in pExo after 24h, 48h of each stage of radiotherapy.PD-L1 mRNA levels in pExo detected at different time points,by using variance analysis of repeated measures design information.Probing the best timing and manner of radiotherapy division which can make PD-L1 express more,guiding clinical practice of radiotherapy combining with immunotherapy.

DETAILED DESCRIPTION:
Radiation therapy can enhance the effect of immunotherapy,but radiation dose and timing are waiting to be solved. At the same time,tissue detection is time-consuming and laborious, liquid biopsy can reflect the information of tumor tissue,PD-L1 mRNA in plasma exosomes (pExo) is expected to be simple, rapid, non-invasive means of detection. The project is planned to explore the consistency analysis of PD-L1 expression level detected in advanced non-small cell cancer patients' cancer tissues and pExo before and after radiotherapy.The investigators have designed five kinds of radiation-division with bioequivalent doses, and detected the expression levels of PD-L1 in pExo after 24h, 48h of each stage of radiotherapy.PD-L1 mRNA levels in pExo detected at different time points,by using variance analysis of repeated measures design information.Probing the best timing and manner of radiotherapy division which can make PD-L1 express more,guiding clinical practice of radiotherapy combining with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological histology and/or cytology confirmed NSCLC;
2. Based on AJCC Cancer Staging, IIIA, IIIB, IV lung cancer patients with NSCLC;
3. PS 0-2;
4. Expected survival > 3 months;
5. Age 18~75 years old;
6. The function of lung, liver, kidney, bone marrow was normal;
7. The patients had not received radiotherapy for previous primary tumor and metastases;
8. At least accept 2-4 cycles of chemotherapy,not disease progression after chemotherapy,start radiotherapy in two weeks after the last cycle of chemotherapy;
9. Wild-type EGFR;
10. Sensitive mutant EGFR, but refused to targeted therapy;
11. In line with the indications of radiotherapy and accept it;
12. Voluntarily enrolled to participate in,better compliance, cooperate with experimental observations, and sign informed consent.

Exclusion Criteria:

1. Vital organs (e.g., heart, liver, kidney) have serious dysfunction;
2. Patients with other malignancies;
3. Patients with a history of autoimmune disease;
4. The patients are pregnant and lactating (Women of childbearing age need to check the pregnancy test);
5. In the activity of acute or chronic infectious diseases;
6. Patients with a clear history of drug allergy or allergic genus;
7. Patients with participating in other clinical trials at the same time;
8. Other cases that researchers believe that patients should not participate in the present trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
The match rate of PD-L1 protein expression in tumor tissue and PD-L1 mRNA expression in pExo before radiotherapy. | up to two and a half years
  The match rate of PD-L1 protein expression in tumor tissue and PD-L1 mRNA
The match rate of PD-L1 protein expression in tumor tissue and PD-L1 mRNA expression in pExo after radiotherapy. | up to two and a half years
  The match rate of PD-L1 protein expression in tumor tissue and PD-L1 mRNA
The best radiotherapy-division which can make PD-L1 express more. | up to two and a half years
  The best radiotherapy-division which can make PD-L1 express more.
The best timing of radiotherapy which can make PD-L1 express more. | up to two and a half years
  The best timing of radiotherapy which can make PD-L1 express more.

SECONDARY OUTCOMES:
Correlation between PD-L1 expression through radiation-induced and the ORR. | up to two and a half years
  Correlation between PD-L1 expression through radiation-induced and the ORR.
Correlation between PD-L1 expression through radiation-induced and the radiation pneumonitis. | up to two and a half years
  Correlation between PD-L1 expression through radiation-induced and the radiation pneumonitis.

CONTACTS AND LOCATIONS:
Overall Officials: jianguo sun, Phd, Study Director — the second affiliated hospital of Army medical university
Locations (1):
- the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality, China